CLINICAL TRIAL: NCT03974776
Title: A PHASE 1, RANDOMIZED, DOUBLE BLIND, SPONSOR-OPEN, PLACEBO-CONTROLLED STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF SINGLE-DOSE, SUBCUTANEOUS ADMINISTRATION OF PF-06946860 TO HEALTHY ADULT JAPANESE PARTICIPANTS
Brief Title: Singe Dose Study of PF- 06946860 in Healthy Adult Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: C3651002; FIP (Other: Alias Study Number); Japanese Ph1 (Other: Alias Study Number)
Record Dates: First submitted 2019-06-03; First posted 2019-06-05 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-06946860 (Experimental): Single subcutaneous administration of PF-06946860
  Interventions: Biological: PF-06946860
- Placebo (Placebo Comparator): Single subcutaneous administration of placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: PF-06946860 — PF-06946860 administered subcutaneously
  Arms: PF-06946860
Other: Placebo — Placebo administered subcutaneously
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of PF-06946860 in healthy adult Japanese participants following single dose administration.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy female subjects of nonchildbearing potential and/or male subjects who, at the time of screening, are between the ages of 18 and 55 years, inclusive
* Body mass index (BMI) within 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb)
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study
* Subjects enrolling as Japanese must have four biologically Japanese grandparents born in Japan.

Key Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing.
* History of allergic reactions to diagnostic or therapeutic protein or human albumin.
* History of recurrent infections or active infection within 28 days of screening.
* Exposure to live vaccines within 28 days of screening.
* History of regular alcohol consumption or positive drug test
* Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of IP (whichever is longer).
* Fertile male subjects who are unwilling or unable to use a highly effective method of contraception for the duration of the study and for at least 28 days after the last dose.
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Incidence of participants experiencing AE | Up to 20 weeks post-dose

SECONDARY OUTCOMES:
Maximum Observed PF-06946860 Concentration (Cmax) | Up to 20 weeks post-dose
Area Under the Curve From Time Zero to Last Quantifiable PF-06946860 Concentration (AUClast) | Up to 20 weeks post-dose
Time to Reach Maximum Observed PF-06946860 Concentration (Tmax) | Up to 20 weeks post-dose
PF-06946860 Half-Life (t1/2) | Up to 20 weeks post-dose, as data permit
  Time measured for the PF-06946860 concentration to decrease by one half.
Incidence of development of ADA, and if necessary NAb, against PF-06946860 | Up to 20 weeks post-dose, as data permit

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Anaheim Clinical Trials LLC-Clinical Research, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3651002